CLINICAL TRIAL: NCT02846350
Title: Positive Connections: COPA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Fundacion Huesped, Buenos Aires, Argentina (Unknown); Fundacion Helios Salud, Buenos Aires, Argentina (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, DEBORAH JONES, Professor of Psychiatry & Behavioral Sciences, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20160313; R01MH095539 (NIH)
Record Dates: First submitted 2016-07-01; First posted 2016-07-27 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV, Motivational Interviewing, Retention in Care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition (Active Comparator): The proposed intervention training utilizes a structured, sustainable MI training and supervision program designed to improve retention, adherence and persistence in challenging patients.
  Interventions: Behavioral: Motivational Interviewing
- Standard of Care (SOC) (No Intervention): Physicians providing SOC will attend 3 time-matched video presentations over 2 years on research on optimizing entry into and retention in care and adherence, from materials available at the International Association for Providers of AIDS Care

INTERVENTIONS:
Behavioral: Motivational Interviewing — The training will include MI skills and elements identified as most effective, MI spirit (collaboration, evoking patient motivation, honoring patient autonomy, recognizing and reinforcing change talk, and "rolling" with (not fighting) resistance. Physicians utilizing MI will learn to engage with patients in an empathic, nonjudgmental manner and to pose simple but strategic questions to motivate change; when patients resist change, the physician learns to ''roll'' with resistance instead of confronting it. If and when the patient is ready to initiate a change, the physician will be prepared to support their decision
  Arms: Experimental condition

SUMMARY:
This study proposes to assess the impact of a provider-based intervention to enhance re-engagement and improve retention, adherence, persistence and viral load among challenging patients in Argentina

DETAILED DESCRIPTION:
Motivational Interviewing (MI) has primarily been utilized as a counseling strategy by therapists to counter addiction and improve lifestyle behaviors.

This application proposes to train physicians to utilize MI to promote re-engagement in HIV care and to sustain retention and adherence. The study will increase the reach of the original pilot study and increase its generalizability, expanding the patient population to a wide variety of public and private clinic and hospital patients, including transgender women, drug users, men who have sex with men (MSM), and heterosexual men and women.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* At least 18 years of age (there will be no upper age range)
* "Challenging" HIV-infected patients, defined as 1) diagnosed for > 6 months and having detectable viral load > 500 copies/mL at last assessment following 6 months of ART prescription, AND 2) not retained in care, i.e., 3 missed pharmacy pick-ups in the last 6 consecutive months, or not attending a physician visit in the last 12 months or more

Exclusion Criteria:

* Participants with delirium and/or psychosis will be excluded.

There are no exclusions based on literacy as all materials will be administered using an audio computer assisted self-interview system (ACASI) supervised by assessors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
HIV viral Load (VL) | Less than 6 months detectable VL
  VL will be assessed by blood sampling. Viral suppression (HIV VL <200 copies/mL) will be the primary dichotomous outcome; a secondary dichotomization will be made among detectable patients with VL <1000 and those with VL >1000.
Retention in care | 2 years
  Defined as the number of missed clinic appointments (i.e., "no shows" not cancelled in advance by patients or clinic staff) in the 6 months preceding assessment.
Medication persistence | 2 years
  Medication persistence is the time to treatment discontinuation, with a permissible gap of < 30 days, participants will be considered to have discontinued the regimen if a therapy gap = > 30 days occurs.
Medication adherence: Hair sample | 2 years
  Adherence by hair sample to estimate an average concentration of ARV medication exposure
Medication adherence: Self-report | 2 years
  Proportion of self-reported adherent participants over time

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Jones, PhD, Principal Investigator — University of Miami
Locations (2):
- Argentina (2):
  - Fundacion Huesped, Buenos Aires
  - Helios Salud, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sued O, Cecchini D, Rolon MJ, Calanni L, David D, Lupo S, Cahn P, Cassetti I, Weiss SM, Alcaide ML, Rodriguez VJ, Mantero A, Jones DL. A small cluster randomised clinical trial to improve health outcomes among Argentine patients disengaged from HIV care. Lancet Reg Health Am. 2022 Sep;13:100307. doi: 10.1016/j.lana.2022.100307. Epub 2022 Jun 23. PMID 36210799
- [Derived] Sued O, Cassetti I, Cecchini D, Cahn P, de Murillo LB, Weiss SM, Mandell LN, Soni M, Jones DL. Physician-delivered motivational interviewing to improve adherence and retention in care among challenging HIV-infected patients in Argentina (COPA2): study protocol for a cluster randomized controlled trial. Trials. 2018 Jul 24;19(1):396. doi: 10.1186/s13063-018-2758-5. PMID 30041703

DOCUMENTS (1):
  • Informed Consent Form (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02846350/ICF_001.pdf